CLINICAL TRIAL: NCT06106256
Title: 3WAVeS: Three-Axis Wearable Adaptive Vestibular Stimulator
Brief Title: Three-Axis Wearable Adaptive Vestibular Stimulator
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gaurav N. Pradhan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23-002124
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the galvanic stimulation (GVS) intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Positive GVS During VR Flight Simulation (Experimental): Subjects will receive positive galvanic vestibular stimulation (GVS) during a flight simulation in virtual reality (VR).
  Interventions: Device: Galvanic Vestibular Stimulation (GVS); Other: Flight simulations in virtual reality (VR)
- Negative GVS During VR Flight Simulation (Experimental): Subjects will receive negative galvanic vestibular stimulation (GVS) during a flight simulation in virtual reality (VR).
  Interventions: Device: Galvanic Vestibular Stimulation (GVS); Other: Flight simulations in virtual reality (VR)
- No GVS During VR Flight Simulation (Experimental): Subjects will not receive any galvanic vestibular stimulation (GVS) during a flight simulation in virtual reality (VR).
  Interventions: Other: Flight simulations in virtual reality (VR)
- Positive GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system (Experimental): Subjects will receive positive galvanic vestibular stimulation (GVS) while utilizing the 3-DOF Bertec Portable Essential's dual-balance force plate system.
  Interventions: Device: Galvanic Vestibular Stimulation (GVS); Other: 3-DOF Bertec Portable Essential's dual-balance force plate system
- Negative GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system (Experimental): Subjects will receive negative galvanic vestibular stimulation (GVS) while utilizing the 3-DOF Bertec Portable Essential's dual-balance force plate system.
  Interventions: Device: Galvanic Vestibular Stimulation (GVS); Other: 3-DOF Bertec Portable Essential's dual-balance force plate system
- No GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system (Experimental): Subjects will not receive any galvanic vestibular stimulation (GVS) while utilizing the 3-DOF Bertec Portable Essential's dual-balance force plate system.
  Interventions: Other: 3-DOF Bertec Portable Essential's dual-balance force plate system

INTERVENTIONS:
Device: Galvanic Vestibular Stimulation (GVS) — Four electrodes, forehead, behind both ears, and back of your neck, provide bidirectional electrical stimulation and receive information about the amplitude delivered accounting for skin impedance
  Arms: Negative GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system; Negative GVS During VR Flight Simulation; Positive GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system; Positive GVS During VR Flight Simulation
Other: Flight simulations in virtual reality (VR) — Highly immersive, 3D virtual flight simulation environment
  Arms: Negative GVS During VR Flight Simulation; No GVS During VR Flight Simulation; Positive GVS During VR Flight Simulation
Other: 3-DOF Bertec Portable Essential's dual-balance force plate system — Firm surface/plate to stand on while being presented disorienting visual patters of moving vertical and/or horizontal bars of alternating black and white.
  Arms: Negative GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system; No GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system; Positive GVS During 3-DOF Bertec Portable Essential's dual-balance force plate system

SUMMARY:
The purpose of this study is to improve current galvanic vestibular stimulation (GVS) technology to ease the motion sickness often associated with virtual reality (VR) simulation.

DETAILED DESCRIPTION:
The Three-Axis Wearable Adaptive Vestibular Stimulator (3WAVeS) technology that combines galvanic vestibular stimulation (GVS) and Virtual Reality (VR) will not only increase VR-based simulation realism and presence, but will also mitigate the motion sickness often associated with VR simulation by re-coupling the vestibular and ocular inputs to the VR user. Additionally, due to GVS technology's ability to accurately provide continuous inputs to the vestibular system, 3WAVeS can intentionally simulate high-fidelity effects of spatial disorientation for training purposes.

ELIGIBILITY:
Inclusion Criteria:

* For our purposes, participants must be able to consent to participate themselves and be 21 to 55 years of age
* Must be able to attend in-person sessions at the Mayo Aerospace Medicine and Vestibular Research Laboratory in Scottsdale, AZ.
* No racial/ethnic groups will be excluded, although all participants must be fluent speakers of English.

Exclusion Criteria:

- History of vestibular disease, migraine, or significant balance disorder; history of severe motion sensitivity, women who are pregnant.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pensacola Diagnostic Index-based motion sickness questionnaire | Immediately after each flight stimulation session, approximately 1 hour
  This index allowed a comparison of motion sickness severity across subjects that may each present with a different constellation of symptoms like nausea, skin color, sweating, salivation, drowsiness, headache, and dizziness. The approach is to have the subject and/or observer grade the subjective intensity of different modalities of symptoms and signs (described below) as slight, moderate or severe. Overall motion sickness severity is then derived from a sum of scores resulting in a weighted "malaise index".
COG Sway velocity | Immediately after balance testing in each session, approximately 1 hour
  The sway angle of the center of gravity (COG) is the measure the amount of sway in any direction. The COG sway velocity is the ratio of the distance traveled by the COG (degrees) to the time (sec) of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Pradhan, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT06106256/ICF_000.pdf